CLINICAL TRIAL: NCT01383746
Title: Efficacy and Tolerance of RADIOEMBOLIZATION for Patients With Unresectable Intrahepatic Cholangiocarcinoma With Tumor Progression After First-line Therapy
Brief Title: Second-line Therapy of Unresectable Cholangiocarcinoma by RADIOEMBOLIZATION
Acronym: CHOLANGIOSIR
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Not enough inclusion
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P100701
Record Dates: First submitted 2011-06-27; First posted 2011-06-28 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2013-08

CONDITIONS: Cholestasis, Progressive Familial Intrahepatic 3
Keywords: Cholangiocarcinoma; RADIOEMBOLIZATION; tumor response; progression-free survival; safety; second-line therapy
MeSH Terms: conditions — Cholestasis, progressive familial intrahepatic 3; Cholangiocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Yttrium microsphere injection
  Interventions: Device: Yttrium microsphere injection

INTERVENTIONS:
Device: Yttrium microsphere injection — Radiation therapy

SUMMARY:
Cholangiocarcinoma (CCK) is a rare tumor (2000 new cases/year in France) with very poor prognosis (overall survival < 3% at 5 years). Less than 20% of patients may benefit from curative surgical resection and most patients have medical treatment by palliative treatment by palliative chemotherapy. It is not standard first-line chemotherapy validated for unresectable CCK, but the best objective response rate (OR) and overall survival (OS) are observed with gemcitabine and platinum associations (OR 24 to 36% and OS between 9.5 to 15.4 months). In case of tumor progression ater this first line therapy, no treatment is currently being validated.

RADIOEMBOLIZATION (RE) is a new, transarterial approach to radiation therapy using 90 Yttrium microspheres.

In the patients with unresectable CCK , the first pilot studies showed interesting results with rates of OR 45 to 90% and a median OS of 14.9 mots and an acceptable safety.

Study Hypothesis : RE could help achieve tumor stabilization in patients with intra-hepatic CCK in tumor progression after first-line therapy.

DETAILED DESCRIPTION:
Extended description of the protocol, including information not already contained in other fields, such as comparison studied.

It is a pilot study including 20 patients with unresectable intra-hepatic CCK in tumor progression after first-line therapy.

Description of the protocol :

1. Information and signed CONSENTMENT
2. Preparatory phase : pre-treatment mesenteric angiography and technetium-99m macroaggregated albumin scans are performed to assess gastrointestinal flow and lung shunting.
3. Therapeutic phase : intra-arterial administration of resin-based microspheres ( SIRSPHERES, SIRTEX). The RE can be performed in 2 sessions, especially if liver disease is bi-lobar.
4. Follow up to J15,M1,M2,M4 and M6 : clinical examination and imaging evaluation ( scans and /or MRI)

ELIGIBILITY:
Inclusion Criteria:

* Unresectable intra-hepatic CCK histologically proven
* Tumor progression documented on imaging evaluation ( CT or MRI) according to RECIST criteria version 1.1 after first-line therapy
* Performance status < 2 ; 4) Bilirubin < 36 micromol/l
* age > 18 years

Exclusion Criteria:

* Extra-hepatic metastases
* Uncontrolled biliary obstruction
* Contra-indications to RE.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2011-10; Primary Completion 2012-08 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Progression -free survival at 6 months (from date of inclusion) | 6 months
  Progression -free survival defined by the number of patients alive at 6 months without tumor progression documented on imaging evaluation ( MRI or CT) using RECIST criteria version 1.1.

SECONDARY OUTCOMES:
Tumor response at 1 month, 2 months, 4 months, 6 months | 1 month, 2 months, 4 months, 6 months
  Tumor response documented on imaging evaluation (MRI or CT) using RECIST criteria version 1.1.
Overall Survival at 6 months | 6 months
Safety of RADIOEMBOLIZATION using the NCI-CTCAE V3.0 classification. | 2 weeks, 1 month, 2 months, 4 months, 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Laetitia FARTOUX, MD,, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hôpital Saint Antoine. Service d'Hépatologie, Pole digestif., Paris, France

REFERENCES:
- [Background] West J, Wood H, Logan RF, Quinn M, Aithal GP. Trends in the incidence of primary liver and biliary tract cancers in England and Wales 1971-2001. Br J Cancer. 2006 Jun 5;94(11):1751-8. doi: 10.1038/sj.bjc.6603127. PMID 16736026
- [Background] Khan SA, Thomas HC, Davidson BR, Taylor-Robinson SD. Cholangiocarcinoma. Lancet. 2005 Oct 8;366(9493):1303-14. doi: 10.1016/S0140-6736(05)67530-7. PMID 16214602
- [Background] Patel T. Increasing incidence and mortality of primary intrahepatic cholangiocarcinoma in the United States. Hepatology. 2001 Jun;33(6):1353-7. doi: 10.1053/jhep.2001.25087. PMID 11391522
- [Background] Gores GJ. Cholangiocarcinoma: current concepts and insights. Hepatology. 2003 May;37(5):961-9. doi: 10.1053/jhep.2003.50200. No abstract available. PMID 12717374
- [Background] Khan SA, Davidson BR, Goldin R, Pereira SP, Rosenberg WM, Taylor-Robinson SD, Thillainayagam AV, Thomas HC, Thursz MR, Wasan H; British Society of Gastroenterology. Guidelines for the diagnosis and treatment of cholangiocarcinoma: consensus document. Gut. 2002 Nov;51 Suppl 6(Suppl 6):VI1-9. doi: 10.1136/gut.51.suppl_6.vi1. No abstract available. PMID 12376491
- [Background] Valle J, Wasan H, Palmer DH, Cunningham D, Anthoney A, Maraveyas A, Madhusudan S, Iveson T, Hughes S, Pereira SP, Roughton M, Bridgewater J; ABC-02 Trial Investigators. Cisplatin plus gemcitabine versus gemcitabine for biliary tract cancer. N Engl J Med. 2010 Apr 8;362(14):1273-81. doi: 10.1056/NEJMoa0908721. PMID 20375404
- [Background] Ducreux M, Van Cutsem E, Van Laethem JL, Gress TM, Jeziorski K, Rougier P, Wagener T, Anak O, Baron B, Nordlinger B; EORTC Gastro Intestinal Tract Cancer Group. A randomised phase II trial of weekly high-dose 5-fluorouracil with and without folinic acid and cisplatin in patients with advanced biliary tract carcinoma: results of the 40955 EORTC trial. Eur J Cancer. 2005 Feb;41(3):398-403. doi: 10.1016/j.ejca.2004.10.026. PMID 15691639
- [Background] Wagner AD, Buechner-Steudel P, Moehler M, Schmalenberg H, Behrens R, Fahlke J, Wein A, Behl S, Kuss O, Kleber G, Fleig WE. Gemcitabine, oxaliplatin and 5-FU in advanced bile duct and gallbladder carcinoma: two parallel, multicentre phase-II trials. Br J Cancer. 2009 Dec 1;101(11):1846-52. doi: 10.1038/sj.bjc.6605377. Epub 2009 Nov 10. PMID 19904267
- [Background] Andre T, Reyes-Vidal JM, Fartoux L, Ross P, Leslie M, Rosmorduc O, Clemens MR, Louvet C, Perez N, Mehmud F, Scheithauer W. Gemcitabine and oxaliplatin in advanced biliary tract carcinoma: a phase II study. Br J Cancer. 2008 Sep 16;99(6):862-7. doi: 10.1038/sj.bjc.6604628. PMID 19238628